CLINICAL TRIAL: NCT01738009
Title: Mechanisms of Pharyngeal Collapse in Sleep Apnea, Study B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David Andrew Wellman, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012P000957B; 1R01HL102321-01A1 (NIH)
Record Dates: First submitted 2012-11-14; First posted 2012-11-30 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Sleep Apnea
Keywords: Sleep Apnea; Pathophysiology
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Induction of flow limitation (Experimental): Flow limitation will be induced by sustained reductions in continuous positive airway pressure during sleep
  Interventions: Other: Induction of flow limitation

INTERVENTIONS:
Other: Induction of flow limitation

SUMMARY:
In obstructive sleep apnea (OSA), the upper airway recurrently closes during sleep. The mechanisms that lead to airway closure are not completely understood. Some studies have shown that there is progressive narrowing of the pharyngeal airway across breaths during expiration (Progressive Expiratory Narrowing, PEN) preceding an obstructive apnea. The cause of PEN is unknown. The investigators will test if lung volumes and low respiratory drive play a role in PEN.

DETAILED DESCRIPTION:
The mechanisms that lead to airway closure in OSA are not completely understood. Some studies have shown that there is progressive narrowing of the pharyngeal airway across breaths during expiration (Progressive Expiratory Narrowing, PEN) preceding an obstructive apnea.

The investigators will test if lung volumes and low respiratory drive play a role in PEN. To this end, the investigators will visualize the pharynx of sleep apnea patients during sleep using a thin endoscope during sleep while simultaneously measuring lung volumes, genioglossus electromyogram, and pharyngeal pressure during flow-limited breaths. Flow limitation will be induced by sustained reductions of continuous positive airway pressure (CPAP).

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects or patients with OSA

Exclusion Criteria:

* Any unstable cardiac condition (other than well controlled hypertension) or pulmonary problems.
* Any medication known to influence breathing, sleep/arousal or muscle physiology
* Concurrent sleep disorders (insomnia, narcolepsy, central sleep apnea or parasomnia)
* Claustrophobia
* Inability to sleep supine
* Allergy to lidocaine or oxymetazoline hydroclhoride
* For women: Pregnancy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-12-08 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Difference in peak inspiratory flow | 3 minutes
  Measured peak inspiratory flow will be compared to predicted peak inspiratory flow during flow restricted breaths.
  The time frame for the outcome will be the duration of induced flow limitation (3 minutes each) . Flow limitation will be induced several times during the night. Flow limited breaths will be averaged.

CONTACTS AND LOCATIONS:
Overall Officials: David A Wellman, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States